CLINICAL TRIAL: NCT06878196
Title: ctDNA-guided First-line Immuno-de-escalation Therapy for Stage IVB and Recurrent Cervical Cancer: A Prospective, Single-arm, Multicenter Phase II Clinical Trial
Brief Title: ctDNA-guided First-line Immuno-de-escalation Therapy for IVB-stage and Recurrent Cervical Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Obstetrics & Gynecology Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FUOBGY-2024-235
Record Dates: First submitted 2025-03-10; First posted 2025-03-14 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Uterine Cervical Neoplasm
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Plasma ctDNA negative group (Experimental): Patients with persistent, recurrent, or advanced metastatic cervical cancer who have not received systemic treatment are treated with cadonilimab combined with cisplatin-based chemotherapy ± bevacizumab (treatment dosage: cadonilimab 10 mg/kg, paclitaxel 175 mg/m^2, cisplatin 50 mg/m^2, cisplatin AUC 4-5, bevacizumab 7.5-15 mg/kg), once every 3 weeks, for a total of 6 cycles (if the patient continues to benefit, chemotherapy is allowed beyond 6 cycles), followed by maintenance treatment with cadonilab ± bevacizumab.During the treatment period, participants undergo a visit for assessment once every 6 weeks.
  Interventions: Drug: cadonilimab combined with cisplatin-based chemotherapy ± bevacizumab

INTERVENTIONS:
Drug: cadonilimab combined with cisplatin-based chemotherapy ± bevacizumab — Patients with persistent, recurrent, or advanced metastatic cervical cancer who have not received systemic treatment are treated with cadonilimab combined with cisplatin-based chemotherapy ± bevacizumab (treatment dosage: cadonilimab 10 mg/kg, paclitaxel 175 mg/m^2, cisplatin 50 mg/m^2, cisplatin AUC 4-5, bevacizumab 7.5-15 mg/kg), once every 3 weeks, for a total of 6 cycles (if the patient continues to benefit, chemotherapy is allowed beyond 6 cycles), followed by maintenance treatment with cadonilab ± bevacizumab.

SUMMARY:
This study aims to evaluate the clinical feasibility of first-line immunochemotherapy for stage IVB and recurrent cervical cancer guided by circulating tumor DNA (ctDNA), in order to explore the optimal treatment duration or criteria for discontinuation of first-line immunotherapy in patients with stage IVB cervical cancer or recurrent cervical cancer. To ensure the quality of the study, before the study begins, the research applicant and participants jointly discuss and formulate the research plan. Necessary steps should be taken during the design and implementation stages of the study to ensure that the collected data is accurate, consistent, complete, and credible.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed as stage IVB primary treatment and recurrent cervical cancer patients (this relapse has not been systematically treated); Histologically or cytologically confirmed recurrent or metastatic cervical cancer, pathological types are squamous cell carcinoma, adenocarcinoma, or adenosquamous carcinoma; Age ≥18 years old and ≤75 years old, female; Signed written informed consent form, and able to comply with the visitation and related procedures specified in the protocol; Has not received systematic treatment for primary stage IVB or this relapse; Has at least one measurable lesion (RECIST 1.1 version); ECOG performance status 0-1; Estimated survival time ≥3 months; Menopausal trial participants must agree to use effective contraceptive measures during the trial; pregnant women must have a negative serum or urine pregnancy test.

Good organ function:

Hematology (subjects will not be allowed to receive blood transfusion or growth factor support within 7 days of starting the study): i. Neutrophil count (ANC) ≥ 1.5 × 10^9 /L (1,500/mm^3); ii. Platelet count ≥ 100 × 10^9 /L (100,000/mm^3); iii. Hemoglobin ≥ 9.0 g/dL.

Kidney:

i. Serum creatinine (SCr) ≤ 1.5 × ULN or creatinine clearance (CrCl) calculated value ≥ 50 mL/min * using the Cockcroft-Gault formula to calculate CrCl; if cisplatin is planned to be used in combination, CrCl ≥ 60 mL/min;

Liver:

i. Serum total bilirubin (TBil) ≤ 1.5 × ULN; for subjects with liver metastasis or with evidence of Gilbert's disease, TBil ≤ 3 × ULN; ii. AST and ALT ≤2.5 × ULN; for subjects with liver metastasis, AST and ALT ≤ 5 × ULN; iii. Serum albumin ≥ 28 g/L.

Coagulation:

i. International normalized ratio and activated partial thromboplastin time ≤ 1.5 × ULN (unless the subject is undergoing anticoagulant treatment, and the coagulation parameters (PT/INR and aPTT) are within the expected range of anticoagulant treatment at screening) 11. Menopausal trial participants must agree to use effective contraceptive measures during the trial; pregnant women must have a negative serum or urine pregnancy test.

Exclusion Criteria:

* Patients with pathological types other than squamous cell carcinoma, adenocarcinoma, or adenosquamous carcinoma (e.g., small cell carcinoma, clear cell carcinoma, etc.).

Patients with clinically significant hydronephrosis of the renal pelvis, judged by the investigator as not relievable by nephrostomy or ureteral stent placement. Presence of central nervous system metastasis or carcinomatous meningitis.

Patients with other active malignant tumors within 3 years prior to the first dose of medication, except for locally curable tumor types that are considered cured, such as cutaneous squamous cell carcinoma, cutaneous basal cell carcinoma, superficial bladder carcinoma, primary breast cancer.

Within 4 weeks prior to the first dose of medication, patients who have received the last cycle of concurrent radiochemotherapy aimed at radical or neoadjuvant/adjuvant purposes; within 2 weeks prior to the first dose of medication, patients who have received palliative radiotherapy (e.g., for bone metastasis); within 2 weeks prior to the first dose of medication, patients who have received drugs with immunomodulatory effects (e.g. thymic peptides, interferons, interleukin-2); within 2 weeks prior to the first dose of medication, patients who have received traditional Chinese patent medicine for anti-tumor adaptation.

Patients who have previously received immune checkpoint inhibitors (e.g., anti PD-1 antibodies, anti PD-L1 antibodies, anti CTLA-4 antibodies, etc.) or any treatment targeting tumor immune mechanisms (e.g., antibodies targeting ICOS, CD40, CD137, GITR, OX40 targets, etc.).

Within 4 weeks prior to the first dose of medication, patients who have undergone major surgery (determined by the investigator), open biopsy, or significant trauma; or patients who require major surgical treatment during the study period and cannot tolerate medication.

Patients with active or potentially recurrent autoimmune diseases; the following are excluded: vitiligo, alopecia, psoriasis, or eczema that do not require systemic treatment; hypothyroidism caused by autoimmune thyroiditis, requiring only stable dose hormone replacement treatment; type I diabetes requiring only stable dose insulin replacement treatment.

Within 14 days prior to the first dose of medication, patients who require systemic treatment with >10 mg/day prednisone or equivalent doses of glucocorticoid hormones or other immunosuppressive drugs; within 4 weeks prior to the first dose of medication, patients with severe infections, including but not limited to complications requiring hospitalization, sepsis, or severe pneumonia.

Active or potentially recurrent systemic infections requiring systemic treatment (including active pulmonary tuberculosis and active syphilis infection), and who have used systemic antibacterial, antiviral, or antifungal drugs within 2 weeks prior to the first dose of medication; note: antiviral drugs for hepatitis B are excluded.

Active hepatitis B virus carriers, non-active or asymptomatic hepatitis B virus (HBV) carriers (hepatitis B surface antigen [HBsAg] positive) with HBV DNA >1000 IU/mL, and active hepatitis C virus carriers (note: non-active or asymptomatic carriers, after treatment and stable hepatitis B carriers with HBV DNA ≤ 1000 IU/mL are allowed to enroll). Patients with cured hepatitis C are allowed to enroll.

Patients with active or a history of inflammatory bowel disease (e.g. Crohn's disease, ulcerative colitis), active diverticulitis, presence of clinical manifestations of gastrointestinal obstruction, or those requiring routine parenteral fluid, parenteral nutrition, or nasogastric tube placement.

Severe cerebrovascular or cerebrovascular diseases. Previous antineoplastic treatment toxicity not resolved, defined as toxicity not recovered to NCI CTCAE v5.0 ≤1 grade, or the levels specified in the inclusion/exclusion criteria (except for alopecia).

Patients allergic to the investigational medication. Any condition that the investigator believes may pose a risk to receiving study medication treatment, or may interfere with the evaluation of the study medication or the safety or interpretation of the results of the study (e.g. patients with other serious diseases or psychiatric disorders, etc.)

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-03-10 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
The accuracy of plasma ctDNA as a guide for adaptive immune chemotherapy in patients with stage IVB and recurrent cervical cancer. | The time frame was from subject enrollment until post-treatment follow-up for two years

CONTACTS AND LOCATIONS:
Locations (1):
- The Obstetrics and Gynecology Hospital of Fudan University, Shanghai, Shanghai Municipality, China